CLINICAL TRIAL: NCT03551574
Title: An Observational Study of Retinal Function and Structure After Repair of Macula-involving Retinal Detachment Complicated by Proliferative Vitreoretinopathy (RDPVR) Using Adaptive Optics
Brief Title: Adaptive Optics in PVR
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CHAD1033
Record Dates: First submitted 2018-05-10; First posted 2018-06-11 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Macular involving retinal detachment: Patients with retinal detachments that have developed PVR when the macula has been involved

SUMMARY:
The purpose of this study is to investigate the loss of retinal cells following retinal detachment surgery using an imaging device called an adaptive optics camera. The retina is a thin layer which lines the back of the eye. It is sensitive to light (like the film in a camera) and is necessary for vision. If a hole or rip develops in a retina it can become detached. The macula is the central portion of the retina which the investigators use for fine vision. This area can also become detached as part of a retinal detachment. Proliferative vitreoretinopathy (PVR) is an abnormal scarring response inside the eye which can occur when the retina detaches. It can adversely affect the outcome of the retinal detachment repair and is associated with a worse visual prognosis. The investigators want to investigate retinal cell loss in patients with retinal detachments that have developed PVR when the macula has been involved.

The investigators plan to compare them to two other groups of patients, who have not developed PVR:

1. Patients with macula-involving retinal detachments without PVR
2. Patients with macula-sparing detachments without PVR

The investigators will investigate retinal cell loss in these types of retinal detachments using adaptive optics imaging. This is a non-invasive imaging technique which allows the investigators to view the retina at very high magnification. Investigating photoreceptor loss and its association with visual outcome in this way should help to guide future interventions in promoting retinal regeneration. The investigators plan to recruit 25 patients at one UK hospital. The project is funded by the charity Fight for Sight.

DETAILED DESCRIPTION:
A cohort of 10 cases of macula-involving retinal detachment complicated by proliferative vitreoretinopathy grade C (RDPVR group) will be identified from vitreoretinal clinics at Moorfields Eye Hospital. 26 weeks following retinal detachment repair, and after removal of any silicone oil tamponade, these cases will undergo post-operative visual assessment, OCT imaging and microperimetry. These investigations will be correlated with adaptive optics (AO) enface imaging of cone photoreceptors at the macula. This will be compared with groups of 10 cases of macula involving retinal detachment without PVR (RD-OFF) and 5 cases of macula-sparing retinal detachment (RD-ON). Both comparison groups (RD-OFF & RD-ON) will undergo assessments at both 6 weeks and 26 weeks post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* RD-PVR group: patients who have had successful retinal surgery to treat macular-involving retinal detachment with PVR C.
* RD-OFF group: patients who have had successful retinal surgery to treat macular-involving retinal detachment without PVR.
* RD-ON group: patients who have had successful retinal surgery to treat macular-sparing retinal detachment without PVR.
* 18 years of age

Exclusion Criteria:

* Media opacity precluding imaging (including silicone oil tamponade)
* Poor central fixation (defined as a fixation score of <10 out of 20)
* Recent contact lens (CLs) wear in the last 48 hours
* Previous refractive surgery/ other corneal surgery
* Spherical equivalent refractive error exceeding -12 or +6D
* Irregularly shaped pupil
* Unable to be dilated
* Unable to give informed consent
* Ocular co-morbidity affecting visual outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with retinal detachments that have developed PVR when the macula has been involved
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
The difference in cone density in patients following repair of macula-involving retinal detachment in eyes with PVR (RD-PVR), versus macula-involving retinal detachment without PVR (RD-OFF) at 26 weeks following retinal detachment repair. | 6 months
  The difference in cone density in patients following repair of macula-involving retinal detachment in eyes with PVR (RD-PVR), versus macula-involving retinal detachment without PVR (RD-OFF) at 26 weeks following retinal detachment repair. Images will be taken with an adaptive optics camera.

SECONDARY OUTCOMES:
Estimate differences in cone mosaics in the PVR-RD vs RD-OFF groups. | 6 months
  Estimate differences in cone mosaics in the PVR-RD vs RD-OFF groups.
Estimate differences in cone mosaics in the PVR-RD & RD-ON groups.3 | 6 months
  Estimate differences in cone mosaics in the PVR-RD & RD-ON groups.
Estimate differences in cone mosaics in the RD-OFF & RD-ON groups | 6 months
  Estimate differences in cone mosaics in the RD-OFF & RD-ON groups
Estimate correlation between cone mosaics and post-operative visual acuity & microperimetry | 6 months
  Estimate correlation between cone mosaics and post-operative visual acuity & microperimetry
Estimate correlation between cone mosaics and retinal layer changes on SD-OCT | 6 months
  Estimate correlation between cone mosaics and retinal layer changes on SD-OCT
Estimate differences in cone mosaics at 6 weeks and 26 weeks following retinal detachment repair (RD-OFF & RD-ON groups only) | 6 months
  Estimate differences in cone mosaics at 6 weeks and 26 weeks following retinal detachment repair (RD-OFF & RDIRAS Estimate differences in cone mosaics at 6 weeks and 26 weeks following retinal detachment repair (RD-OFF & RD-ON groups only)
Exploratory correlation comparison between visual function variables in PVR patients, and various matrices of cone mosaic from AOC | 6 months
  Exploratory correlation comparison between visual function variables in PVR patients, and various matrices of cone mosaic from AOC

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom